CLINICAL TRIAL: NCT03718442
Title: Low Energy Dissection Vs. Electrocautery Qualitative Severity and Depth of Thermal Artifact in Breast Cancer Lumpectomy Shaved Surgical Margins
Brief Title: Low Energy Dissection Vs. Electrocautery in Lumpectomy Shaved Surgical Margins
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Invuity, Inc. (Industry)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-8984
Record Dates: First submitted 2018-10-18; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue - Shaved margins for cancer detection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Breast cancer patients - lumpectomy: Women who are 18 years or older, have Ductal carcinoma in situ (DCIS) or invasive breast-conserving surgery, have not had previous chest radiotherapy. 20 patients who meet above study population criteria will be enrolled in this study.Shaved margins for each lumpectomy site will be excised with either Bovie (3 sides) or PhotonBlade (3 sides) for each patient. The effect of PhotonBlade vs Bovie on pathology assessment of lumpectomy shaved surgical margins will be compared.
  Interventions: Device: PhotonBlade vs Bovie for lumpectomy shaved surgical margins

INTERVENTIONS:
Device: PhotonBlade vs Bovie for lumpectomy shaved surgical margins — For each enrolled patient, six shaved margins will be obtained (superior, inferior, medial, lateral, anterior, and posterior). For each patient, electrocautery will be used to obtain 3 of the shaved margins, and PhotonBlade to obtain the other 3 shaved margins. Once the lumpectomy site shaved margins have been obtained, the shaved surgical margins will be evaluated by a pathologist whom is blinded in regards to the dissection device that was used for each margin. The pathologist will be evaluating each shaved margin and reporting the outcomes (qualitative severity and depth of thermal artifact)

SUMMARY:
The purpose of this study is to compare the qualitative severity and depth of dissection devices' associated thermal artifact in breast lumpectomy shaved margins between the use of electrocautery and low thermal energy dissection, PhotonBlade.

The investigators hypothesize that the use of PhotonBlade would result in a significantly lower qualitative severity and a shorter depth of thermal artifact in breast lumpectomies shaved margins, when compared to electrocautery devices.

DETAILED DESCRIPTION:
When performing lumpectomy, surgeons have used electrocautery devices as dissecting tools. However, those devices use high thermal energy that might impact the margin cellular architecture and as such the quality of margin assessment by the pathologist. Moreover, recently, modern low thermal energy dissection devices have been introduced to the market. However, the impact of those devices on reducing the thermal injury/artifact on surgical margin has not been well investigated. 4,5 While Ruidaz et al. 2011 data suggest that using the traditional electrosurgical device in place of the low thermal-injury device results in 48% of the close margin samples being negatively converted to false-positive, and in 11% converting from close to false-negative, there is still a need for more studies to further characterize the utility of those devices. 6 PhotonBlade (Invuity, San Francisco, CA, USA) has been approved by United States Food and Drug Administration (FDA). PhotonBlade is a dynamic precision illuminator with enhanced energy delivery dissection device. The dynamic precision illumination is a thermally cool illumination technology that allows a uniformal illumination without glare or shadow. 7 The enhanced energy delivery technology allows low thermal spread, surgeon controlled edge temperature, and wet field use.7 As such, PhontonBlade allows better blade control for achieving adequate visualization, hemostasis, with a minimum collateral damage to the surgical margin tissue. The use of PhotonBlade demonstrated the least penetrating thermal tissue damage/spread when compared to other modern dissection devices (Valleylab Pencil, Valleylab EDGE Coated Pencil, PlasmaBlade 3.0S and PlasmaBlade 4.0).8

ELIGIBILITY:
Inclusion Criteria:

* have aged 18 years old or older.
* have DCIS or Invasive breast cancer that is eligible for breast-conserving surgery.
* have not had previous chest radiotherapy.
* understand the study purpose, requirements, and risks.
* able and willing to give informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer in women
Study Population: Women who have a diagnosis of breast cancer and undergo a lumpectomy
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Severity of thermal artifact | Through study completion, an average of 6 months
  The severity of the thermal artifact will be assessed by identifying the presence or absence of each the three qualitative severity zones, described previously,6 as below:
  * Zone I: extensive charring tissue
  * Zone II: fused cellular architecture
  * Zone III: distressed cellular architecture
Depth of thermal artifact | Through study completion, an average of 6 months
  The depth of the thermal artifact will be assessed by reporting the length in micrometer (μm) from the start of Zone 1 to the end of Zone III.

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place at this time.

REFERENCES:
- [Background] ACS. Breast Cancer Facts and Figures 2011-2012. (2012).
- [Background] Vila J, Gandini S, Gentilini O. Overall survival according to type of surgery in young (</=40 years) early breast cancer patients: A systematic meta-analysis comparing breast-conserving surgery versus mastectomy. Breast. 2015 Jun;24(3):175-81. doi: 10.1016/j.breast.2015.02.002. Epub 2015 Feb 23. PMID 25728282
- [Background] Pleijhuis RG, Graafland M, de Vries J, Bart J, de Jong JS, van Dam GM. Obtaining adequate surgical margins in breast-conserving therapy for patients with early-stage breast cancer: current modalities and future directions. Ann Surg Oncol. 2009 Oct;16(10):2717-30. doi: 10.1245/s10434-009-0609-z. Epub 2009 Jul 17. PMID 19609829
- [Background] Chiappa C, Rovera F, Corben AD, Fachinetti A, De Berardinis V, Marchionini V, Rausei S, Boni L, Dionigi G, Dionigi R. Surgical margins in breast conservation. Int J Surg. 2013;11 Suppl 1:S69-72. doi: 10.1016/S1743-9191(13)60021-7. PMID 24380558
- [Background] Ruidiaz ME, Cortes-Mateos MJ, Sandoval S, Martin DT, Wang-Rodriguez J, Hasteh F, Wallace A, Vose JG, Kummel AC, Blair SL. Quantitative comparison of surgical margin histology following excision with traditional electrosurgery and a low-thermal-injury dissection device. J Surg Oncol. 2011 Dec;104(7):746-54. doi: 10.1002/jso.22012. Epub 2011 Jul 8. PMID 21744349
- [Background] Haydon E. et al. Assessment of penetrating thermal tissue damage/spread associated with PhotonBlade™, Valleylab™ Pencil, Valleylab™ EDGE™ Coated Pencil, PlasmaBlade® 3.0S and PlasmaBlade® 4.0 for intraoperative tissue dissection using the fresh extirpated porcine muscle model